CLINICAL TRIAL: NCT02997644
Title: The Effect of an Educational Pain Approach Before Elective Lower-extremity Surgery on 6-month Post-operative Use of Opioid Medication: A Randomized Clinical Trial
Brief Title: Impact of Different Educational Approaches on Post-operative Opiate Utilization After Elective Lower Extremity Surgery
Acronym: OpiateLEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dan Rhon, Senior Scientist, Center for the Intrepid, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C.2016.142d
Record Dates: First submitted 2016-12-06; First posted 2016-12-20 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Knee Injuries and Disorders; Hip Injuries and Disorders; Opiate Addiction
Keywords: patient education; orthopaedic surgery; post-surgical pain; chronic opioid use
MeSH Terms: conditions — Knee Injuries; Disease; Hip Injuries; Opioid-Related Disorders; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video Education (Experimental): Video education delivered on a tablet computer
  Interventions: Behavioral: Video Education
- Usual Care Group (Placebo Comparator): Regular information about opioid usage they typically receive from their surgeon.
  Interventions: Behavioral: Usual Care Group

INTERVENTIONS:
Behavioral: Video Education — The content of the education focuses on providing a historical perspective for opioid prescription from the time when the risk of dependence was highly underestimated. The video discusses the current evidence for the effect of opioid medications in non-cancer non-acute pain. It also discusses some of the dangers of long-term opioid usage.
  The consent, enrollment, and video education will take about 20-30 minutes for patients in this group, and occur at the end of their preoperative visit. The patient will watch the video on a portable Tablet computer.
  Arms: Video Education
Behavioral: Usual Care Group — Patients that are randomized to usual care will only receive the regular instructions about opioid usage they typically receive from their surgeon.
  Arms: Usual Care Group

SUMMARY:
The purpose of this study is to evaluate the use of post-operative opioid use after two different educational interventions. The investigators will compare changes in pain, disability and sleep between groups 6 months after elective lower extremity surgery.

DETAILED DESCRIPTION:
Hypothesis: The primary hypothesis is that the educational intervention provided prior to the surgery and prior to the prescription, will result in a greater understanding and awareness of the deleterious effects of long-term use of opioid based medications, and in turn reduce utilization post-operatively in the long-term (6 months).

Specific Aim 1: Evaluate prescription opioid medication use for the 6-month period after surgery in subjects that received the education compared to those that received usual care education.

Specific Aim 2: Compare the changes in self-reported outcome measures (pain, disability, and sleep) between groups over the 6-month period after surgery.

Specific Aim 3: Describe the sociodemographic factors and healthcare utilization in enrolled subjects for the 12 months leading up to a surgical procedure. Identify factors that could account for differences in opioid medication utilization, and any potential interaction effect between intervention, opioid use, and clinical outcomes following surgery.

Study Procedures/Research Interventions:

Subjects will be randomized to either receive usual care only or usual care plus the education video. Usual care is defined as typical information the surgeon would otherwise provide the patient before surgery. All patients will receive the usual care education from their surgeon.

Randomization:

Subjects will then be randomized into one of two arms (Group I = Educational Video, Group II= Usual Care Only). The method of group assignment will be sequentially numbered opaque sealed envelopes (SNOSE). To minimize the risk of predicting the treatment assignment of the next eligible patient, randomization will be performed in permuted blocks of two or four with random variation of the blocking number.

All Subjects:

All subjects will receive the usual care education that is typically given by their surgeon. That will be left up to the discretion of each surgeon. The screening and enrollment should take no more than 5-10 minutes, and then the filling out of self-report questionnaires should take approximately 5-7 minutes. Subjects in the group that is randomized to the education will take an additional 11 minutes to view the educational content.

All patients will proceed with the surgical procedure as planned. Each week during the 1-month period after the surgery, patients will be contacted (phone call, email, and text message - depending on what they consented to).

At the 1-month and 6-month time points they will be asked to fill out the additional clinical outcomes measures detailed below. These can be done in person with a visit to the clinic or over the telephone.

Sample Size Estimation. Collection of healthcare utilization will occur in 100% of the subjects as no follow-up is required, and therefore no opportunities to collect data from a follow-up visit will be lost. A sample of 120 subjects should allow us to determine significant differences between groups, based on a moderate effect size of 0.6.

ELIGIBILITY:
Inclusion Criteria:

1. Any Tricare-eligible patient scheduled for a pre-operative surgery appointment for an elective orthopaedic surgery of the hip, knee, or foot/ankle at SAMMC.
2. The surgery is taking place for a condition that has been ongoing for 6 months or longer (chronic)
3. Between the age of 18 - 65 years
4. Read and speak English well enough to understand the education, provide informed consent and follow study instructions (the surgeon, investigators, or research assistants will make this determination. Any patient that needs an interpreter will not be allowed to enroll).

Exclusion Criteria:

1. Known aversion or allergy that would prevent the patient from taking any opioid-based pain medication (any contraindications to using opioids)
2. History of prior surgery to the same location.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Opiate Prescriptions | 6 months
  Total opiate prescriptions

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | baseline, 1 month, 6 months
  A 0-10 numeric pain rating scale ('0' indicating no pain, and '10' worst imaginable pain) will be used to assess LBP intensity. Numeric pain scales are known to have excellent test-retest reliability.
PROMIS-29 | baseline, 1 month, 6 months
  The Patient Reported Outcomes Measurement Information Systems (PROMIS) 29-item short form (version 2) to assess disability. The PROMIS 29-item short form efficiently assesses several outcomes important to patients with a neuromusculoskeletal injury, including pain intensity and interference, sleep disturbance, anxiety, depression, fatigue, and social role participation using items developed with rigorous methodology and patient input. The PROMIS-29 scores have been found valid for patients with orthopedic injuries, with minimum clinically important change thresholds of 2-4 points for most scales. It has also been used to successfully measure psychosocial resiliency in patients with disability.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rhon, DSc, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing must go through a Data Sharing Agreement via the Defense Health Agency
Time Frame: Usually 1 year, but agreement is contract-specific with the Defense Health Agency
Access Criteria: Submit a Data Sharing Agreement Application through the DHA
URL: https://www.health.mil/Military-Health-Topics/Privacy-and-Civil-Liberties/Submit-a-Data-Sharing-Application

REFERENCES:
- [Background] French MT, McGeary KA, Chitwood DD, McCoy CB. Chronic illicit drug use, health services utilization and the cost of medical care. Soc Sci Med. 2000 Jun;50(12):1703-13. doi: 10.1016/s0277-9536(99)00411-6. PMID 10798326
- [Background] Songer TJ, LaPorte RE. Disabilities due to injury in the military. Am J Prev Med. 2000 Apr;18(3 Suppl):33-40. doi: 10.1016/s0749-3797(00)00107-0. PMID 10736539
- [Background] Vanderlip ER, Sullivan MD, Edlund MJ, Martin BC, Fortney J, Austen M, Williams JS, Hudson T. National study of discontinuation of long-term opioid therapy among veterans. Pain. 2014 Dec;155(12):2673-2679. doi: 10.1016/j.pain.2014.09.034. Epub 2014 Sep 30. PMID 25277462
- [Background] Toblin RL, Quartana PJ, Riviere LA, Walper KC, Hoge CW. Chronic pain and opioid use in US soldiers after combat deployment. JAMA Intern Med. 2014 Aug;174(8):1400-1. doi: 10.1001/jamainternmed.2014.2726. No abstract available. PMID 24978399
- [Background] Rozet I, Nishio I, Robbertze R, Rotter D, Chansky H, Hernandez AV. Prolonged opioid use after knee arthroscopy in military veterans. Anesth Analg. 2014 Aug;119(2):454-459. doi: 10.1213/ANE.0000000000000292. PMID 24977636
- [Background] Dobscha SK, Morasco BJ, Duckart JP, Macey T, Deyo RA. Correlates of prescription opioid initiation and long-term opioid use in veterans with persistent pain. Clin J Pain. 2013 Feb;29(2):102-8. doi: 10.1097/AJP.0b013e3182490bdb. PMID 23269280
- [Derived] Rhon DI, Greenlee TA, Mayhew R, Boyer C, Laugesen M, Roth J, Dowd TC, Gill NW. Engaging Education About Risks of Opioid Use With Patients Before Elective Surgery of the Lower Extremity Did Not Reduce Postoperative Opioid Utilization: A Randomized Controlled Trial. J Am Acad Orthop Surg. 2022 Apr 1;30(7):e649-e657. doi: 10.5435/JAAOS-D-21-00603. PMID 35130200